CLINICAL TRIAL: NCT02702869
Title: Allied Cleft & Craniofacial Quality-Improvement and Research Network (ACCQUIREnet): Prospective Data-collection System and Learning Health-care Network for the Comprehensive Appraisal of Cleft and Craniofacial Care
Brief Title: Allied Cleft & Craniofacial Quality-Improvement and Research Network (ACCQUIREnet)
Acronym: ACCQUIREnet
Status: Enrolling by invitation | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00104806
Record Dates: First submitted 2015-10-16; First posted 2016-03-09 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cleft Lip; Cleft Palate; Cleft Lip and Palate
Keywords: cleft lip; cleft palate; cleft lip and palate; cleft alveolus; multidisciplinary team; interdisciplinary team
MeSH Terms: conditions — Cleft Lip; Cleft Palate | interventions — Sphincterotomy, Transduodenal; Orthognathic Surgery; Rhinoplasty; Middle Ear Ventilation; Speech Therapy; Orthodontics; Nasoalveolar Molding; Audiometry; Hearing Aids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 22 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- uCL(A): Children with unilateral cleft lip with/without cleft alveolus but intact secondary palate. Subgroup analysis by severity of lip (complete, incomplete, or lesser-form).
  Interventions: Procedure: cleft lip repair; Procedure: gingivoperiosteoplasty; Procedure: LeFort-1 maxillary repositioning; Procedure: rhinoplasty; Other: speech therapy; Procedure: orthodontia; Procedure: presurgical orthopedics
- uCL(A)P: Children with unilateral cleft lip with/without cleft alveolus and with cleft secondary palate. Subgroup analysis by severity of lip (complete, incomplete, or lesser-form) and severity of palate (submucous, Veau-I, Veau-II, or Veau-III).
  Interventions: Procedure: cleft lip repair; Procedure: cleft palate repair; Procedure: oronasal fistula repair; Procedure: pharyngoplasty; Procedure: gingivoperiosteoplasty; Procedure: LeFort-1 maxillary repositioning; Procedure: rhinoplasty; Procedure: myringotomy and tympanostomy tube placement; Other: speech therapy; Procedure: orthodontia; Procedure: presurgical orthopedics; Device: sound amplification for hearing
- bCL(A): Children with bilateral cleft lip with/without cleft alveolus but intact secondary palate. Subgroup analysis by severity of lip (complete, incomplete, or lesser-form).
  Interventions: Procedure: cleft lip repair; Procedure: gingivoperiosteoplasty; Procedure: LeFort-1 maxillary repositioning; Procedure: rhinoplasty; Other: speech therapy; Procedure: orthodontia; Procedure: presurgical orthopedics
- bCL(A)P: Children with unilateral cleft lip with/without cleft alveolus and with cleft secondary palate. Subgroup analysis by severity of lip (complete, incomplete, or lesser-form) and severity of palate (submucous, Veau-I, Veau-II, Veau-III, or Veau-IV).
  Interventions: Procedure: cleft lip repair; Procedure: cleft palate repair; Procedure: oronasal fistula repair; Procedure: pharyngoplasty; Procedure: gingivoperiosteoplasty; Procedure: LeFort-1 maxillary repositioning; Procedure: rhinoplasty; Procedure: myringotomy and tympanostomy tube placement; Other: speech therapy; Procedure: orthodontia; Procedure: presurgical orthopedics; Device: sound amplification for hearing
- CP: Children with cleft secondary palate only, but intact lip and alveolus. Subgroup analysis by severity (submucous, Veau-I, or Veau-II).
  Interventions: Procedure: cleft palate repair; Procedure: oronasal fistula repair; Procedure: pharyngoplasty; Procedure: LeFort-1 maxillary repositioning; Procedure: myringotomy and tympanostomy tube placement; Other: speech therapy; Device: sound amplification for hearing

INTERVENTIONS:
Procedure: cleft lip repair
  Other Names: cheiloplasty
  Groups: bCL(A); bCL(A)P; uCL(A); uCL(A)P
Procedure: cleft palate repair
  Other Names: palatoplasty
  Groups: CP; bCL(A)P; uCL(A)P
Procedure: oronasal fistula repair
  Groups: CP; bCL(A)P; uCL(A)P
Procedure: pharyngoplasty
  Other Names: sphincteroplasty
  Groups: CP; bCL(A)P; uCL(A)P
Procedure: gingivoperiosteoplasty
  Groups: bCL(A); bCL(A)P; uCL(A); uCL(A)P
Procedure: LeFort-1 maxillary repositioning
  Other Names: orthognathic surgery
Procedure: rhinoplasty
  Groups: bCL(A); bCL(A)P; uCL(A); uCL(A)P
Procedure: myringotomy and tympanostomy tube placement
  Groups: CP; bCL(A)P; uCL(A)P
Other: speech therapy
Procedure: orthodontia
  Groups: bCL(A); bCL(A)P; uCL(A); uCL(A)P
Procedure: presurgical orthopedics
  Other Names: nasoalveolar molding; dentofacial orthopedics; Georgiade-Latham appliance; Latham appliance
  Groups: bCL(A); bCL(A)P; uCL(A); uCL(A)P
Device: sound amplification for hearing
  Other Names: hearing aid
  Groups: CP; bCL(A)P; uCL(A)P

SUMMARY:
The Allied Cleft & Craniofacial Quality-Improvement and Research Network (ACCQUIREnet) is a group of multidisciplinary cleft teams that have implemented a system for prospective collection of outcomes data, based on the ICHOM Standard Set for the Comprehensive Appraisal of Cleft Care, CLEFT-Q, and other outcomes instruments. Participating cleft teams may analyze clinical and psychosocial outcomes related to care of the child with cleft lip and/or palate (CL/P), compare its performance with those of other cleft centers, and identify opportunities for quality improvement.

DETAILED DESCRIPTION:
The purpose of this project is to implement a system of prospective, standardized data collection for all patients with cleft lip and/or palate (CL/P) treated by the cleft and craniofacial centers that participate in ACCQUIREnet.

Adoption of this prospective data-collection system has two principal goals:

1. To enable on-demand and scheduled review of cleft-care-related safety and outcomes data and team performance for the purpose of internal audits and continuous quality improvement; and
2. To permit participation in multi-site, collaborative quality-improvement projects and/or research networks that require usage of these standardized data-collection methods. (These collaborations are described in corresponding IRB protocols and data-transfer agreements. Patient privacy and confidentiality is protected at all times.)

All patients with CL/P treated at cleft and craniofacial centers participating in ACCQUIREnet will be invited to participate in this project. Duke University serves as the coordinating center and statistical support center for the study. Data are maintained in a local, secured database.

The IRB protocol details methods of quality assurance, data monitoring, and auditing. Data dictionaries employed in ACCQUIREnet include the CleftCap REDCap project template, CleftKit Common Data Model (an extension of the PCORnet Common Data Model), the ICHOM Standard Set for the Comprehensive Appraisal of Cleft Care, and the CLEFT-Q patient-reported outcome manual, maintained by the International Consortium for Health Outcomes Measurement (ichom.org) and McMaster University, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Typical orofacial clefts, of which subtypes are:
* Unilateral or bilateral cleft lip
* Unilateral or bilateral cleft lip and alveolus
* Unilateral or bilateral cleft lip and alveolus and palate
* Unilateral or bilateral cleft lip and palate
* Overt cleft palate
* Occult cleft palate

Exclusion Criteria:

* Atypical (Tessier) facial clefts

Ages: 1 Day to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients born with cleft lip and/or palate are eligible for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Speech: intelligibility | ~5 years of age
  Utilizes the intelligibility in context scale (ICS)
Speech: intelligibility | ~8 years of age
  Utilizes the intelligibility in context scale (ICS)
Speech: intelligibility | ~12 years of age
  Utilizes the intelligibility in context scale (ICS)
Speech: intelligibility | ~22 years of age
  Utilizes the intelligibility in context scale (ICS)
Speech: velopharyngeal competence | ~5 years of age
Speech: velopharyngeal competence | ~8 years of age
Speech: velopharyngeal competence | ~12 years of age
Speech: velopharyngeal competence | ~22 years of age
Speech: articulation | ~5 years of age
  Utilizes the modified percent correct consonants (mPCC) scale
Speech: articulation | ~8 years of age
  Utilizes the modified percent correct consonants (mPCC) scale
Speech: articulation | ~12 years of age
  Utilizes the modified percent correct consonants (mPCC) scale
Speech: articulation | ~22 years of age
  Utilizes the modified percent correct consonants (mPCC) scale
Speech: patient-reported outcomes related to speech and speaking | ~8 years of age
  Utilizes the CLEFT-Q PROM
Speech: patient-reported outcomes related to speech and speaking | ~12 years of age
  Utilizes the CLEFT-Q PROM
Speech: patient-reported outcomes related to speech and speaking | ~22 years of age
  Utilizes the CLEFT-Q PROM
Hearing: puretone average | ~5 years of age
Dental: dmft and DMFT scores | ~5 years of age
  Utilizes the dmft score for deciduous teeth and DMFT score for permanent teeth
Dental: dmft and DMFT scores | ~12 years of age
  Utilizes the dmft score for deciduous teeth and DMFT score for permanent teeth
Dental: dmft and DMFT scores | ~22 years of age
  Utilizes the dmft score for deciduous teeth and DMFT score for permanent teeth
Dental: occlusion (Uses modifications of the GOSLON scale) | ~5 years of age
Dental: occlusion (Uses modifications of the Bauru scale) | ~5 years of age
Dental: occlusion (Uses modifications of the GOSLON scale) | ~12 years of age
Dental: occlusion (Uses modifications of the Bauru scale) | ~12 years of age
Dental: occlusion (Uses modifications of the GOSLON scale) | ~22 years of age
Dental: occlusion (Uses modifications of the Bauru scale) | ~22 years of age
Dental: patient-reported outcomes related to mastication | ~8 years of age
  Uses the CLEFT-Q PROM
Dental: patient-reported outcomes related to mastication | ~12 years of age
  Uses the CLEFT-Q PROM
Dental: patient-reported outcomes related to mastication | ~22 years of age
  Uses the CLEFT-Q PROM
Dental: patient-reported outcomes related to oral health | ~8 years of age
  Uses the COHIP PROM
Dental: patient-reported outcomes related to oral health | ~12 years of age
  Uses the COHIP PROM
Dental: patient-reported outcomes related to oral health | ~22 years of age
  Uses the COHIP PROM
Patient-reported outcomes related to eating/drinking | ~8 years of age
  Uses the CLEFT-Q PROM
Patient-reported outcomes related to eating/drinking | ~12 years of age
  Uses the CLEFT-Q PROM
Patient-reported outcomes related to eating/drinking | ~22 years of age
  Uses the CLEFT-Q PROM
Breathing: Patient-reported outcomes related to nasal and oral breathing | ~8 years of age
  Uses the NOSE PROM
Breathing: Patient-reported outcomes related to nasal and oral breathing | ~12 years of age
  Uses the NOSE PROM
Breathing: Patient-reported outcomes related to nasal and oral breathing | ~22 years of age
  Uses the NOSE PROM
Aesthetics: Patient-reported outcomes related to appearance | ~8 years of age
  Uses the CLEFT-Q PROM
Aesthetics: Patient-reported outcomes related to appearance | ~12 years of age
  Uses the CLEFT-Q PROM
Aesthetics: Patient-reported outcomes related to appearance | ~22 years of age
  Uses the CLEFT-Q PROM
Aesthetics: Clinical assessment of nasolabial and facial aesthetics | ~2 years of age
Aesthetics: Clinical assessment of nasolabial and facial aesthetics | ~5 years of age
Aesthetics: Clinical assessment of nasolabial and facial aesthetics | ~8 years of age
Aesthetics: Clinical assessment of nasolabial and facial aesthetics | ~12 years of age
Aesthetics: Clinical assessment of nasolabial and facial aesthetics | ~22 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Allori, MD, MPH, Principal Investigator — Duke University
Locations (11):
- United States (10):
  - University of Florida - Shands Hospital, Gainesville, Florida
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Orlando Health - Arnold Palmer Hospital for Children, Orlando, Florida
  - Johns Hopkins - All Children's Hospital (JHACH), St. Petersburg, Florida
  - Maine Medical Center, Portland, Maine
  - Harvard University - Boston Children's Hospital (BCH), Boston, Massachusetts
  - Washington University - St. Louis Children's Hospital (WUSTL), St Louis, Missouri
  - Duke University - Duke Children's Hospital & Health Center, Durham, North Carolina
  - Wake Forest University - Brenner Children's Hospital, Winston-Salem, North Carolina
  - University of Texas at Houston - Children's Memorial Hermann Hospital, Houston, Texas
- Dalhousie University - IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
This is a collaborative research network. All data processing happens at the coordinating center, with results reviewed by the participating centers.

REFERENCES:
- See also: Duke Cleft & Craniofacial Center — https://www.dukehealth.org/pediatric-treatments/pediatric-plastic-and-reconstructive-surgery/cleft-lip-and-cleft-palate
- See also: Official web site for ICHOM Standard Set for cleft lip and/or palate, upon which the Duke project is based — http://www.ichom.org/medical-conditions/cleft-lip-palate/
- See also: ACCQUIREnet web site — http://accquire.net